CLINICAL TRIAL: NCT05983094
Title: Study of Utidelone Based Neoadjuvant Treatment on Early High-risk or Locally Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); First Affiliated Hospital of China Medical University (Unknown)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of the Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4047
Record Dates: First submitted 2023-07-18; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Epirubicin; Trastuzumab; pertuzumab

STUDY DESIGN:
Intervention Model Description: Study of Utidelone based neoadjuvant treatment on early high-risk or locally advanced breast cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cohort 1 Triple-negative breast cancer (Experimental): Hormone Receptor(HR) negative, Human Epidermal Growth Factor Receptor 2(HER2 )negative breast cancer Drug: Utidelone in combination with carboplatin Utidelone injection 30mg/m2, on days 1-5 of each cycle; Carboplatin ,Area Under Curve(AUC)6, iv, was administered on day 1; One treatment cycle is 21 days, and there are 6 cycles in total.
  Interventions: Drug: Utidelone; Drug: Carboplatin
- cohort 2 HR positive, HER2 negative breast cancer (Experimental): HR positive, HER2 negative, Immunohistochemical(IHC)0,1+; 2+, Fluorescence in situ hybridization(FISH)non-amplification breast cancer Drug: Utidelone in combination with Epirubicin Utidelone injection 30mg/m2, on days 1-5 of each cycle; Epirubicin 75mg/m2 was administered on day 1; One treatment cycle is 21 days, and there are 6 cycles in total.
  Interventions: Drug: Utidelone; Drug: Epirubicin
- cohort 3 HER2 positive (IHC 3+; IHC 2+,FISH amplification) breast cancer (Experimental): Drug: Utidelone in combination with carboplatin, trastuzumab and pertuzumab Utidelone injection 30mg/m2, on days 1-5 of each cycle; Carboplatin Area Under Curve(AUC)6, iv, was administered on day 1; One treatment cycle is 21 days, and there are 6 cycles in total. Trastuzumab 8mg/kg iv in first cycle on day 1, then 8mg/kg in the rest cycles; pertuzumab 840mg/kg iv in first cycle on day 1, then 420mg/kg in the rest cycles.
  One treatment cycle is 21 days, and there are 6 cycles in total.
  Interventions: Drug: Utidelone; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Utidelone — Utidelone injection 30mg/m2, on days 1-5 of each cycle
Drug: Carboplatin — Carboplatin Area under curve(AUC)6, iv, was administered on day 1
  Arms: cohort 1 Triple-negative breast cancer; cohort 3 HER2 positive (IHC 3+; IHC 2+,FISH amplification) breast cancer
Drug: Epirubicin — Epirubicin 75mg/m2 was administered on day 1
  Arms: cohort 2 HR positive, HER2 negative breast cancer
Drug: Trastuzumab — Trastuzumab 8mg/kg iv in first cycle on day 1, then 6mg/kg in the rest cycles
  Arms: cohort 3 HER2 positive (IHC 3+; IHC 2+,FISH amplification) breast cancer
Drug: Pertuzumab — Pertuzumab 840mg/kg iv in first cycle on day 1, then 420mg/kg in the rest cycles
  Arms: cohort 3 HER2 positive (IHC 3+; IHC 2+,FISH amplification) breast cancer

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Utidelone based regimen as neoadjuvant treatment With High-risk Early-stage or Locally Advanced Breast Cancer.

DETAILED DESCRIPTION:
This is a single arm, multi-center study,three-cohort, prospective phase II study which will enroll 181 high-risk early-stage or locally advanced breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients who will receive initial treatment, 18-70 years of age；
2. Newly diagnosed high-risk early stage (T1c-2, N1; T2, N0) and locally advanced (T1c-2, N2-3; T3-4, N0-3) breast cancer (tumor stage II, III), in which HR+/HER2- T2, N0 patients need to be accompanied by high-risk factors (histological grade 3 or Ki67 ≥ 20%). Triple negative breast cancer(TNBC), HER2 positive (Immunohistochemical(IHC)3+; IHC 2+, FISH amplification) breast cancer, HR negative HER2 IHC 2+ and undetermined result of FISH, HR positive HER2 negative (IHC 0,1+; 2+, FISH amplification) breast cancer confirmed by pathological test.
3. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1
4. The blood routine examination was basically normal (CTCAE ≤ 1) within one week before enrollment (based on the normal values of each research center laboratory). No Human Granulocyte Colony Stimulating Factor(rhGCSF) or blood transfusion/erythropoietin(EPO) or other drugs were used within 14 days prior to enrollment.

   White blood cell count (WBC) ≥ 4 x109 / L; Neutrophil count (ANC) > 1.5x109 / L; Platelet count (PLT) ≥ 100×109/L Hemoglobin(Hb) ≥ 100g/L.
5. The blood biochemistry examination was basically normal (CTCAE ≤ 1) within one week before enrollment (based on the normal values of each research center laboratory) Serum total bilirubin ≤ Upper limit of normal value(ULN)； Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 1.5×ULN； Alkaline phosphatase ≤ 2.5×ULN； Serum creatinine ≤ 1.5×ULN.
6. Color Doppler echocardiography left ventricular Ejection fraction (LVEF) ≥ 55%
7. Female patients with fertility must agree to use effective contraceptive methods during the study period and within 6 months of the last study medication. The Pregnancy test (urine or serum) must be negative
8. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Primary stage IV breast cancer；
2. Inflammatory breast cancer;
3. Bilateral primary breast cancer (including invasive cancer and carcinoma in situ)；
4. Previous anti-cancer treatment or radiotherapy for any malignant tumor, excluding cured cervical Carcinoma in situ, skin Basal-cell carcinoma and squamous cell carcinoma.
5. Receive any sex hormone treatment (such as contraceptives, ovarian hormone replacement therapy, etc.), except for Ovarian function suppression（OFS）fertility protection, or any hormone drugs (such as Raloxifene, tamoxifen, or other selective estrogen receptor modulators) to treat osteoporosis or prevent breast cancer；
6. The patient has undergone major surgery unrelated to breast cancer within 4 weeks before treatment or has not yet fully recovered;
7. Symptomatic peripheral neuropathy CTCAE 5.0 grade ≥ 2
8. Serious cardio cerebral Vascular disease, including but not limited to the followings:
9. History of congestive heart failure or systolic dysfunction (LVEF<50%);
10. Angina pectoris requiring anti angina drugs;
11. High risk uncontrolled arrhythmias or severe conduction abnormalities, such as ventricular arrhythmias that require clinical intervention, II-III degree atrioventricular block, etc; Under resting state, the average corrected Q-T interval(QTcF) of three 12 lead electrocardiogram examinations is>470ms;
12. Clinically significant heart valve disease with cardiac dysfunction;
13. Hypertension that cannot be controlled;
14. History of myocardial infarction
15. Allergic to any component of any drug in this protocol.
16. Those who are not suitable for using Corticosteroid.
17. Individuals with active infections who currently require systematic anti infection treatment.
18. History of immune deficiency disease, including positive of HIV/AIDS, or other acquired or congenital immune deficiency diseases, or having a history of organ transplantation.
19. Who had participated in other drug intervention clinical trials within the 28 days of randomization, or who is participating in another clinical trial or is using other investigational treatments.
20. Individuals in pregnancy (positive Pregnancy test) and lactation.
21. Any other comorbidities that interfere with the implementation of the treatment plan, or the researcher evaluate that the subject has a history of other serious systemic diseases, or other reasons lead to the patients is unsuitable to participate in this trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (etpCR, Pathologic staging after neoadjuvant therapy(yp)T0/is, (yp)N0) | 24 months
  Percentage of patients with absence of invasive neoplastic cells in ipsilateral lymph nodes and breast

SECONDARY OUTCOMES:
Breast Pathologic Complete Response ((bpCR, Pathologic staging after neoadjuvant therapy(yp)T0/is) | 24 months
  Percentage of patients whose pathological evaluation of hematoxylin and eosin-stained breast samples do not show any residual invasive carcinoma
Event Free Survival(EFS) of 2 years | 24 months
  Time from the first dose of study intervention administration to any of the following events: progression of disease that precludes surgery, local or distant recurrence after surgery, second primary malignancy (breast or other invasive cancers), or death due to any cause.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion，an average of 1 year
  Graded according to the Common Terminology Criteria for Adverse Event (CTCAE) grade and changes in CTCAE grade
Patient reported outcome (PRO) | Through study completion，an average of 1 year
  National Cancer Center of China-Breast Cancer-A 1.0 (NCC-BC-A 1.0) during the study was used to assess the quality of life；The minimum to maximum values: 0 , 100 Meaning: the higher scores mean a better outcome.
Patient reported outcome (PRO) | Through study completion，an average of 1 year
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-chemotherapy-induced peripheral neuropathy(CIPN) twenty-item scale (QLQ-CIPN20) was used to assess the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China